CLINICAL TRIAL: NCT07308444
Title: Validation of a Risk Matrix for Severe Postdischarge Pain After Ambulatory Gynaecological Laparoscopy
Brief Title: Predicting Pain After Ambulatory Gynaecological Laparoscopies
Acronym: POP-Matrix
Status: Enrolling by invitation | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marlin Comelon, Senior Physician, Anesthesiologist, PhD, Oslo University Hospital
Other Study IDs: 939735
Record Dates: First submitted 2025-12-05; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Pain
Keywords: Risk matrix
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As day surgery is increasingly preferred over in-hospital treatment due to feasibility and reduced economic costs, it is important to evaluate patient-related outcomes such as comfort and safety after discharge. Most previous studies on predictors for postoperative pain have not focused on postdischarge pain. In a previous study, we found that over 42% of the patients experienced severe postdischarge pain within the first 24 h after ambulatory gynaecologocal laparoscopic surgery, that is a pain score of 7-10 on the NRS. We identified four preoperative risk factors independently associated with severe postdischarge pain. We have developed a risk matrix to predict who will suffer from severe pain after surgery. The risk matrix needs to be validated in a new gynaecological patient sample. It has the potential to improve clinical practice by providing clinicians with a simple, evidence-based tool that can identify high-risk patients before surgery. The scoring takes less than one minute. Today, we do not have such an instrument at hand. The results from this project could influence current routines and treatments at Oslo University Hospital and may also apply to other patient populations and other hospitals.

The primary research objective is to validate a previously developed risk matrix for postdischarge pain in gynecological day-surgery patients.

DETAILED DESCRIPTION:
Early identification of patients at high risk for severe pain can contribute to better and more targeted individual pain prevention and management, thereby reducing the incidence of unnecessary pain and discomfort after surgery. By identifying and treating patients who are particularly vulnerable to severe postoperative pain, we can also reduce the length of hospital stays, prevent unplanned admissions due to pain, decrease the number of outpatient inquiries related to pain, and expedite recovery and return to normal activities. This will contribute to reduced resource use, improved patient care, and hopefully increased patient satisfaction.

In this prospective observational cohort study, we will collect post-discharge pain data necessary to validate a previously developed risk matrix at two different time points: T1) preoperatively on the day of surgery, and T2) during a follow-up call on POD1. In addition, patients' postoperative pain will be assessed using the NRS during PACU stay.

According to the sample size calculation (n=188) + at least 10%, we will include at least 207 patients.

There is no risk connected to participation in the study. All patients will receive standard medical and surgical treatment throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years of age at the time of signing the informed consent.
2. Participant scheduled for ambulatory gynaecological laparoscopy.
3. Capable of giving written informed consent.
4. Must speak and read Norwegian.

Exclusion Criteria:

1. Severe psychiatric disorder, severe cognitive dysfunction.
2. Intraoperative ketamine or lidocaine infusion or regional anaesthesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women by biological sex
Study Population: Women scheduled for ambulatory gynaecological laparoscopic procedures such as: ovarian cyst removal, excision of endometriosis, salpingo-oophorectomy, salpingectomy, chromopertubation, ovarian drilling for polycystic ovary syndrome, adhesion removal, diagnostic laparoscopy, oophorectomy, removal of migrated intrauterine device, sterilisation/tubal ligation.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Severe postdischarge pain | Time from hospital discharge until 24 hours after end of surgery.
  Numerical rating scale for pain, severe pain defined as 7-10 on scale.

SECONDARY OUTCOMES:
Preoperative use of opioids | Last four weeks prior to surgery
Age | Age in years at time for surgery
Preoperative pain | At time for surgery
  Patient NRS (0-10) level before surgery
Pain expectation | After surgery
  Expected postoperative pain intensity (NRS 0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT07308444/Prot_SAP_000.pdf